CLINICAL TRIAL: NCT06765408
Title: The Effect of Facial Yoga on Tonus, Stiffness and Elasticity of Mimic Muscles
Brief Title: Effect of Face Yoga on Mimic Muscles
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hazel Çelik Güzel, Assist. Prof. Dr., Bandırma Onyedi Eylül University
Other Study IDs: 2024 -113
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Facial Yoga; Facial Exercises
Keywords: facial yoga; Myoton; tonus; stiffness; elasticity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: facial yoga exercise program — An exercise programme consisting of basic yoga movements such as swan neck exercise, fist exercise, hand to head exercise, jowl drawer exercise, tongue and palate exercise, lip curling exercise, ceiling kissing exercise, namaste exercise, balloon inflation, spider and fish exercise, lip spray, Chinese moustache, binocular exercise, gaze exercises and lion pose was applied. Each session was approximately 30 minutes and all exercises were accompanied by breathing exercises on the basis of exercising all facial muscles. The exercise programme was performed for 8 weeks, 2 days a week face-to-face and 5 days at home, for a total of 16 sessions face-to-face and 40 sessions at home. Participants were given verbal, written and video explanations and instructions about the exercise protocol. Every day in a WhatsApp group where all participants take part, Assist. Prof. Dr. Hazel Çelik Güzel provided information and reminders and ensured the continuity of the exercises. Participants were al

SUMMARY:
This study aimed to investigate the effect of facial yoga on tonus, stiffness and elasticity of facial muscles.

DETAILED DESCRIPTION:
This study was conducted on healthy volunteers aged 25-50 between June 2024 and January 2025. In the participants who agree to participate in the study, a descriptive data form and myotone evaluations of facial muscles will be performed. Measurements will be carried out immediately after the participants are recruited and at the end of the 8-week facial yoga programme.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 25-50 years of age whose voluntary consent was obtained

Exclusion Criteria:

* Botox application to the facial area in the last 6 months,
* Regular use of analgesics and anti-inflammatories,
* The presence of infection or tumoural structures within the structures in the facial region,
* With TMJ disc displacement and joint degeneration,
* Cervical or TMJ fracture, systemic disease, musculoskeletal problem with evidence of specific pathological condition,
* Any surgical operation related to cervical or TMJ problem,
* Less than 6 months of cervical or TMJ-related physiotherapy and rehabilitation services,
* The one with facial paralysis,
* Participants with diagnosed psychiatric illness will not be included in the study.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The female gender is eligible to participate.
Study Population: Healthy female volunteers
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the mimic muscles tone | June 2024- August 2024
  Myoton®PRO (Myoton Ltd, Myoton AS, Estonia) was used to objectively evaluate of the participants' facial muscles tone. The frontalis, corrugator supercili, orbicularis oculi, nasalis, orbicularis oris, mentalis and buccinator muscles, as well as masseter, temporal and digastric muscles were evaluated bilaterally in the sitting position.
Evaluation of the mimic muscles stiffness | June 2024- August 2024
  Myoton®PRO (Myoton Ltd, Myoton AS, Estonia) was used to objectively evaluate of the participants' facial muscles stiffness. The frontalis, corrugator supercili, orbicularis oculi, nasalis, orbicularis oris, mentalis and buccinator muscles, as well as masseter, temporal and digastric muscles were evaluated bilaterally in the sitting position.
Evaluation of the mimic muscles elasticity | June 2024- August 2024
  Myoton®PRO (Myoton Ltd, Myoton AS, Estonia) was used to objectively evaluate of the participants' facial muscles elasticity. The frontalis, corrugator supercili, orbicularis oculi, nasalis, orbicularis oris, mentalis and buccinator muscles, as well as masseter, temporal and digastric muscles were evaluated bilaterally in the sitting position.

SECONDARY OUTCOMES:
Assessing mimic muscle tone after exercising | October 2024- December 2024
  After the exercise program, the participants' facial muscles tone evaluated by Myoton Pro. The frontalis, corrugator supercili, orbicularis oculi, nasalis, orbicularis oris, mentalis and buccinator muscles, as well as masseter, temporal and digastric muscles were evaluated bilaterally in the sitting position.
Assessing mimic muscle stiffness after exercising | October 2024- December 2024
  After the exercise program, the participants' facial muscles stiffness evaluated by Myoton Pro. The frontalis, corrugator supercili, orbicularis oculi, nasalis, orbicularis oris, mentalis and buccinator muscles, as well as masseter, temporal and digastric muscles were evaluated bilaterally in the sitting position.
Assessing mimic muscle elasticity after exercising | October 2024- December 2024
  After the exercise program, the participants' facial muscles elasticity evaluated by Myoton Pro. The frontalis, corrugator supercili, orbicularis oculi, nasalis, orbicularis oris, mentalis and buccinator muscles, as well as masseter, temporal and digastric muscles were evaluated bilaterally in the sitting position.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided